CLINICAL TRIAL: NCT04230304
Title: A Phase II Study of Daratumumab and Ibrutinib for Relapsed / Refractory Chronic Lymphocytic Leukemia Treatment (DIRECT)
Brief Title: Daratumumab and Ibrutinib for the Treatment of Relapsed or Refractory Chronic Lymphocytic Leukemia, DIRECT Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1784; NCI-2020-00010 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1784 (Other: Mayo Clinic in Florida); 19-001475 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — daratumumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (daratumumab, ibrutinib) (Experimental): Patients receive daratumumab IV on days 1, 8, 15, and 22 of cycles 1-2, on days 1 and 15 of cycles 3-6, and then on day 1 of subsequent cycles. Beginning in cycle 2, patients also receive ibrutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab; Drug: Ibrutinib

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765

SUMMARY:
This phase II trial studies how well daratumumab and ibrutinib work in treating patients with chronic lymphocytic leukemia that has come back (relapsed) or has not responded to previous treatment (refractory). Daratumumab is a monoclonal antibody which works with the body's immune system to destroy cancer cells. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving daratumumab and ibrutinib may work better in treating patients with chronic lymphocytic leukemia compared to ibrutinib alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall response rate after 6 cycles of treatment with daratumumab in combination with ibrutinib in patients who are on /or are previously treated with ibrutinib. (Cohort 1) II. Determine the overall response rate after 6 cycles of treatment with daratumumab in combination with ibrutinib in patients who are naive to ibrutinib treatment. (Cohort 2)

SECONDARY OBJECTIVES:

I. Determine the best overall response rate to treatment with daratumumab plus ibrutinib at any time during the course of the therapy. (Cohort 1) II. The overall incidence of MRD (minimal residual disease) negative state and the time to achieving MRD negativity at any time during this therapy. (Cohort 1) III. Progression free survival (as determined by the International Workshop on Chronic Lymphocytic Leukemia [IWCLL] criteria) among all patients. (Cohort 1) IV. The overall toxicity profile of daratumumab/ibrutinib treatment in this group of patients. (Cohort 1) V. Determine the best overall response rate to treatment with daratumumab plus ibrutinib at any time during the course of the therapy. (Cohort 2) VI. The overall incidence of MRD (minimal residual disease) negative state and the time to achieving MRD negativity at any time during this therapy. (Cohort 2) VII. The overall toxicity profile of daratumumab/ibrutinib treatment in this group of patients. (Cohort 2)

OUTLINE:

Patients receive daratumumab intravenously (IV) on days 1, 8, 15, and 22 of cycles 1-2, on days 1 and 15 of cycles 3-6, and then on day 1 of subsequent cycles. Beginning in cycle 2, patients also receive ibrutinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study registration, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-CLL, confirmed by flow cytometry and as per the criteria outlined by the IWCLL/Hallek December 2008
* Patients must have relapse or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) who have received at least 1 prior anti-CLL/SLL therapy. (Note: There is no upper limit of how many lines of therapy the patient may have received previously)

  * Note: For the purpose of a particular therapy/regimen to be counted towards the number of prior treatments a patient must have received at least 2 cycles of the regimen e.g., a patient who change their treatment regimen after only 1 cycle (due to toxicity or any other reason) will not be considered to have "2" prior therapies
* Patients on low dose prednisone (≤ 10 mg) for treatment of conditions other than CLL are eligible
* Cohort 1 only: Exposed to previous bruton tyrosine kinase (BTK) inhibitor. Patients must meet one of the following criteria:

  * They have been previously treated with a previous BTK inhibitor and were taken off for any reason (except grade 4 toxicity definitely attributed to BTK inhibitor) as long as deemed safe by the treatment physician to receive ibrutinib
  * Currently on a BTK inhibitor and now have progressive disease (BTK inhibitor refractory)
  * Currently on BTK inhibitor and have failed to achieve either a complete remission after at least 12 cycles of treatment with BTK or have suboptimal response (< partial response [PR]) after being on BTK inhibitor treatment for 6 cycles
* Patients must have a measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 at registration
* Absolute neutrophil count >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Hemoglobin >= 7 g/dl (obtained =< 14 days prior to registration)
* Platelets >= 50,000/mm^3 (obtained =< 14 days prior to registration)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) *OR* creatinine clearance > 25 ml/min) (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 mg/dL or direct bilirubin =< 1.0 mg/dL for patients with Gilbert's syndrome (obtained =< 14 days prior to registration)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN (obtained =< 14 days prior to registration)
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 3 months after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug
* Negative pregnancy test done =< 14 days prior to registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Patient is known to have chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal (Note: FEV1 testing is required for subjects suspected of having chronic obstructive pulmonary disease and subjects must be excluded if FEV1 < 50% of predicted normal)
* Patient is known to have moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification (Note: subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study)
* Since this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown, any of the following will deem the subject ineligible for the study:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Patients who have received no prior therapy for CLL
* Patients with history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix, unless in complete remission and off therapy for that disease for > 3 years)
* Patients who have previously received daratumumab or any other anti-CD38 therapy on a clinical trial or for any other malignancy
* Prior or current exposure to any of the following:

  * Exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer.
  * Focal radiation therapy within 14 days prior to randomization with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with a strong cytochrome P450 modulators (CYP3A inhibitor and/or CYP3A inducers). NOTE: A comprehensive list of inhibitors, inducers, and substrates may be found at http://medicine.iupui.edu/clinpharm/ddis/main-table/.
* Major surgery =< 4 weeks prior to registration
* Patients who are:

  * Seropositive for human immunodeficiency virus (HIV)
  * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
  * Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)
* Clinically significant cardiac disease, including:

  * Myocardial infarction within 6 months before randomization, or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
  * Uncontrolled cardiac arrhythmia
  * Screening 12-lead ECG showing a baseline corrected QT interval (QTc) >40 msec.
* Known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins, Dara SC or its excipients (refer to the IB) or known sensitivity to mammalian-derived products
* Have received vaccination with live attenuated vaccines within 4 weeks of first study agent administration
* Patients with inability to swallow capsules or tablets, or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption (malabsorption syndrome, resection of the small bowel, poorly controlled inflammatory bowel disease, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2025-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Previous BTK Inihibitor Exposed); Cohort 2 (BTK Inihibitor naïve): Patients receive daratumumab IV on days 1, 8, 15, and 22 of cycles 1-2, on days 1 and 15 of cycles 3-6, and then on day 1 of subsequent cycles. Beginning in cycle 2, patients also receive ibrutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort 1 (Previous BTK Inihibitor Exposed) | Cohort 2 (BTK Inihibitor naïve)
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Previous BTK Inihibitor Exposed) | Cohort 2 (BTK Inihibitor naïve) | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (4.68) | 60.5 (0.71) | 66.6 (5.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate by Cycle 7
Description: Will be evaluated in each cohort independently. A response is defined as an objective status of complete response (CR), CR with incomplete marrow recovery (CRi), complete clinical response (CCR), nodular partial response (nPR), or PR after 6 cycles of combination treatment. In each cohort, the proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent exact binomial confidence intervals for the true success proportion will be calculated.
Time Frame: 7 months
Population: Both cohorts are analyzed together to avoid deidentifying the outcome for individual patents. Neither arm has enough patients to represent a valid estimate for overall response rate. These results should not be used to compare this treatment to any other treatment or to compare patient cohorts. These results are only reported for regulation purposes. Both cohorts are analyzed together to avoid deidentifying the outcome for the two cohort B patents.
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (Daratumumab, Ibrutinib)
Number analyzed (Participants) | 8
proportion of participants | 0.375

2. Secondary Outcome: Overall Response Rate
Description: Will be evaluated in each cohort independently. Will be estimated by the number of patients who achieve a CR, CRi, CCR, nPR, or PR at any time during combination treatment divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success rate will be calculated.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-01

3. Secondary Outcome: Minimal Residual Disease (MRD) Response Rate
Description: Will be evaluated in each cohort independently. Will be estimated by the number of patients who achieve MRD negative response in both blood and bone marrow at any time during combination treatment divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success rate will be calculated. In patients who achieve MRD negative response, time to achieve MRD negative response will be summarized descriptively (median, range). Time to achieve MRD negative response is defined as time from registration to the earliest date of documentation of MRD negative response in both blood and bone marrow.
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Progression-free Survival
Description: Will be evaluated in each cohort independently. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Adverse Events
Description: Will be evaluated in each cohort independently. Platelets and hemoglobin will be graded according to the Grading Scale for Hematologic Adverse Events in Chronic Lymphocytic Leukemia (CLL) Studies. The maximum grade for each type of adverse event, regardless of causality, will be recorded and reported for each patient, and frequency tables will be reviewed to determine adverse event patterns.
Time Frame: Up to 30 days after completion of study treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 3 years and mortality is still being followed.
Description: Due to lack of accrual, adverse events and morality is reported by treatment group and not cohort. With only two patients accrued to cohort B, it would be unethical to report their isolated adverse events and mortality.
Arm/Group | Treatment (Daratumumab, Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Daratumumab, Ibrutinib) (N=8)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Daratumumab, Ibrutinib) (N=8)
Anemia (Blood and lymphatic system disorders) | 6 (50)
Atrial fibrillation (Cardiac disorders) | 1 (5)
Fatigue (General disorders) | 5 (61)
Bruising (Injury, poisoning and procedural complications) | 6 (133)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (3)
Lymphocyte count increased (Investigations) | 3 (44)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 4 (43)
White blood cell decreased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (19)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT04230304/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT04230304/ICF_001.pdf